CLINICAL TRIAL: NCT04335253
Title: Phase I/IIa First-In-Human Study of EOS884448 in Participants with Advanced Cancers.
Brief Title: First-In-Human Study of EOS884448 in Participants with Advanced Cancers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: iTeos Therapeutics (Industry)
Collaborators: iTeos Belgium SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IO-002
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-09

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multiple Ascending Dose (Experimental): Dose escalation according to cohort allocation
  Interventions: Drug: EOS884448

INTERVENTIONS:
Drug: EOS884448 — Multiple Ascending Dose
  Other Names: EOS-448

SUMMARY:
IO-002 study is a multicenter, open-label, dose-escalation Phase I/IIa clinical study to evaluate the safety and tolerability, PK, PD, and antitumor activity of EOS884448 in participants with advanced cancers.

DETAILED DESCRIPTION:
Multicenter, open-label, dose-escalation Phase I/IIa clinical study to evaluate the safety and tolerability, PK, PD, and antitumor activity of EOS884448 in participants with advanced cancers. The study will consist in a dose-escalation phase to determine the MTD, the RP2D, and the safety of EOS884448 in participants with advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing to provide a signed written informed consent for the trial and consent for biopsies before and during administration of EOS884448
2. Be more than18 years of age on day of signing informed consent.
3. Have histologically or cytologically confirmed advanced or metastatic cancer for whom no standard treatment is further available
4. Have evaluable disease, per RECIST v1.1 for solid tumor escalation or other criteria if indicated
5. Have an ECOG performance status of Grade 0 to 1.
6. Have adequate organ function.
7. Agree to use adequate contraception during the treatment if required.

Exclusion Criteria:

1. Has received any anti-cancer therapy, unless at least 4 weeks (or 5 half-lives, whichever is shorter) since the last dose.
2. Has undergone major surgery within 5 weeks before initiating treatment.
3. Has received prior radiotherapy within 2 weeks of start of IP.
4. Has toxicity (except for alopecia) related to prior anti-cancer therapy, unless the toxicity is resolved, returned to baseline or Grade 1, or deemed irreversible.
5. Has known CNS metastases.
6. Has any condition requiring concurrent use of systemic immunosuppressants or corticosteroids.
7. Has uncontrolled or significant cardiovascular disease.
8. Has received vaccine containing live virus within 4 weeks.
9. Has known active or chronic viral hepatitis.
10. Has any known or underlying medical, psychiatric condition, and/or social situations that, in the opinion of the investigator, would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with Adverse Events | From first dose date to 90 days after the last dose (up to 48 weeks)
Percentage of participants who experience a Dose Limiting Toxicity | From first study treatment administration through Day 28
Define the recommended Phase 2 dose (RP2D) of EOS884448 in participants with advanced tumors. | up to 48 weeks

SECONDARY OUTCOMES:
Mean and median Area under the curve (AUC) of EOS884448 at each dose level | up to 48 weeks
Mean and median Maximum concentration (Cmax) of EOS884448 at each dose level | up to 48 weeks
Percentage of participants with Objective Response as determined by Investigator according to RECIST v1.1or per other specific response criteria according to their tumor type. | From study enrollment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 48 weeks)
Percentage of participants with anti-drug antibodies to EOS884448 | Recorded at baseline (screening), during the first 4 cycles of treatment (4 months), at end of treatment, and 30 and 90 days post last dose (approximately 48 weeks)

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - GZA Ziekenhuizen campus Sint-Augustinus, Antwerp
  - Institut Jules Bordet, Brussels
  - Cliniques universitaires St Luc-UCL, Brussels
  - Universitair Ziekenhuis Gent, Ghent

IPD SHARING:
Plan to Share IPD: No